CLINICAL TRIAL: NCT00684437
Title: Literacy and Smoking Risk Communications
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2006-0699; 1R01CA125413-01 (NIH); NCI-2015-00727 (Registry Identifier: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Smoking
Keywords: Health Literacy; Smoking Risk; Focus Group; Questionnaire; Survey
MeSH Terms: conditions — Smoking | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Factual Gain-Framed (Experimental): Smoking Risk Message - Factual Gain-Framed (FGF)
  Interventions: Behavioral: Focus Group; Behavioral: Questionnaire
- Factual Loss-Framed (Experimental): Smoking Risk Message - Factual Loss-Framed (FLF)
  Interventions: Behavioral: Focus Group; Behavioral: Questionnaire
- Emotional Gain-Framed (Experimental): Smoking Risk Message - Emotional Gain-Framed (EGF)
  Interventions: Behavioral: Focus Group; Behavioral: Questionnaire
- Emotional Loss-Framed (Experimental): Smoking Risk Message - Emotional Loss-Framed (ELF)
  Interventions: Behavioral: Focus Group; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Focus Group — Focus group discussion and evaluation of various smoking risk informational messages. The focus group session should last about 1 hour and 30 minutes.
Behavioral: Questionnaire — Questionnaires taking 15-30 minutes to complete.
  Other Names: Survey

SUMMARY:
Objectives:

Smokers with varying levels of health literacy as assessed by the S-TOFHLA (i.e., inadequate, marginal, adequate) recruited from the community will listen to one of 4 different types of messages emphasizing the health consequences of smoking recorded on a computer in the form of audio scripts (i.e., a human voice pre-recorded on a computer will read each message). Messages written at a 5th to 6th grade reading level will be concurrently presented in written form via a computer monitor and be manipulated in terms of 1) emotionality (i.e., primarily fact- vs. primarily emotion-based), and 2) framing (i.e., gain-framed messages that highlight the potential benefits of quitting smoking vs. loss-framed messages that emphasize the potential costs of failing to quit smoking). Emotionality and framing will be completely crossed to create four different types of messages, 1) factual gain-framed (FGF), 2) factual loss-framed (FLF), 3) emotional gain-framed (EGF), and 4) emotional loss-framed (ELF).

The primary objectives are to:

1. Examine whether main effects emerge for health literacy as assessed by the S-TOFHLA (inadequate, marginal, adequate) and the different message types (fact- vs. emotion-based and gain- vs. loss-framed) on the primary explicit and implicit outcomes: a) intention to quit, and b) implicit and explicit attitudes toward smoking.
2. Examine whether health literacy interacts with the different types of messages (fact-based vs. emotion-based and gain-framed vs. loss-framed) to influence the primary explicit and implicit outcome measures: a) intention to quit smoking, and b) implicit and explicit attitudes toward smoking.

   A secondary, exploratory aim is to:
3. Examine potential associations between a) the primary explicit and implicit outcomes, and b) the secondary explicit and implicit outcomes: knowledge, risk perception, attitudes, self-efficacy, message evaluations, implicit fear of disease, and implicit associations between smoking and disease.

DETAILED DESCRIPTION:
Focus Groups:

If you agree to take part in this study, you will be asked to complete some questionnaires. The questionnaires will ask about your age, income level, education level, and smoking history. This information will allow researchers to look at whether these factors affect how people understand smoking health risk information. The questionnaires will take about 15 minutes to complete. You will also complete a breath test. To complete the breath test, you will blow into a tube that's attached to a machine about the size of a pocket computer. The breath test is used to estimate the amount of tobacco smoke that you inhale.

You will participate in a focus group. During the focus group, research staff will be present to help discuss and evaluate various smoking risk informational messages. You will be asked to decide which messages may be most influential in terms of helping smokers to quit smoking. The messages will include information about health risks of smoking, such as smoking-related cancers, heart disease, lung disease, gum disease, fertility problems, and other related topics.

The focus group session should last about 1 hour and 30 minutes.

The messages will then be selected by the study doctor and used to create pamphlets on the risks of smoking. These pamphlets will be used to help people quit smoking.

Your participation on this study will be over once you have finished taking part in the focus group. All focus groups will be audiotaped and the tape will be sent to an outside company to be transcribed. No information that could be used to identify you such as your name or date of birth will be provided to the outside company.

This is an investigational study. Up to 30 smokers will participate in the focus groups. All will be enrolled at M. D. Anderson.

Pilot Testing and Main Study:

Many people can get and understand smoking health risk information. This study will look at which types of smoking risk information may be most easily understood by different people. Participants in this study will be asked to listen to and read 1 of 4 types of messages on a computer. These messages will talk about and list some health consequences of smoking.

If you agree to take part in this study, you will be asked to complete several questionnaires. These questionnaires will ask about your feelings and moods, thoughts about smoking, risks of smoking, smoking history, and basic information, such as your age, education level, and income level. The questionnaires will take about 30 minutes to complete. You will also complete a breath test. To complete the breath test, you will blow into a tube that's attached to a machine about the size of a pocket computer. The breath test is used to estimate the amount of tobacco smoke that you inhale.

After you have completed these questionnaires and the breath test, you will complete several computer-aided tasks. These computer-aided tasks will allow you to be able to read and hear informational messages about health risks of smoking, such as smoking-related cancers, heart disease, lung disease, gum disease, fertility problems, and other related topics. During this study visit, you will also evaluate several recently designed informational messages on the health risks of smoking. The computer-aided tasks and the evaluation should last about 30 minutes.

After evaluating these messages, you will be asked to complete additional questionnaires in order for researchers to evaluate your responses to them. These questionnaires will ask your opinion about the informational messages and the risks of smoking. These last set of questionnaires should take about 30 minutes to complete. Your participation will be over in this study once you complete the last set of questionnaires.

This is an investigational study. Up to 420 smokers will participate in this part of the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 70 years
2. current smoker with a history of at least 5 cigarettes/day for the last year
3. can speak, read, and write in English
4. home address and a functioning home telephone number

Exclusion Criteria:

1. current use of nicotine replacement therapy or bupropion
2. current enrollment in a smoking cessation treatment program
3. expired CO<10 ppm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2008-05-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Factors that may influence how smokers understand smoking health risk informational messages. | 2 years
  Examine whether main effects emerge for health literacy as assessed by the Short Test of Functional Health Literacy in Adults (S-TOFHLA) (inadequate, marginal, adequate) and the different message types (fact- vs. emotion-based and gain- vs. loss-framed) on the primary explicit and implicit outcomes: a) intention to quit, and b) implicit and explicit attitudes toward smoking

CONTACTS AND LOCATIONS:
Overall Officials: Lorna H. McNeill, MPH,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org